CLINICAL TRIAL: NCT00536055
Title: Dyadic Coping in Breast and Prostate Cancer Patients and Their Spouses - A Pilot Stdy
Brief Title: Dyadic Coping in Breast and Prostate Cancer Patients and Their Spouses
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Herzog Hospital (Other)
Other Study IDs: TASMC - 07 - BC-07309
Record Dates: First submitted 2007-09-26; First posted 2007-09-27 (Estimated); Last update posted 2007-09-27 (Estimated); Status verified 2007-09

CONDITIONS: Breast Cancer; Prostate Cancer; Dyadic Coping
Keywords: breast cancer; prostate cancer; dyadic coping
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to focus on dyadic coping as one of the main factors that enhance resilience in adjustment to cancer, while also assessing other protective factors for coping with traumatic events.

Specifically, the study aims are:

1. To assess the level of post traumatic distress, functional impairment and depression among breast and prostate cancer patients and their spouses.
2. To assess resiliency factors such as flexibility, self efficacy and ego resilience among breast and prostate cancer patients and their spouses.
3. To examine the pattern of dyadic coping at 3 time points: at the beginning and end of radiation therapy, and at six-week follow-up.
4. To examine the relationships between dyadic coping and level of posttraumatic distress and the resilience factors over time (in 3 repeated measures) Different aspects of coping with the trauma of cancer and its treatment may be assessed. Measures of strength and distress amongst patients and their spouses may enable a fuller picture of what types of responses exist, which interventions may be most beneficial, and what other factors may relate to positive coping, increased resilience and quality of life, such as flexibility, and the nature of the couples' dyadic coping.

DETAILED DESCRIPTION:
Introduction:

In the proposed study, we will investigate the risk and protective factors for healthy coping amongst breast and prostrate cancer patients and their spouses. A special focus will be on dyadic coping patterns, i.e. how do the coping patterns of the patient and his/her spouse correlate and how does the spousal response facilitate or impede the outcome of coping of the patient.

Different aspects of coping with the trauma of cancer and its treatment may be assessed. Measures of strength and distress amongst patients and their spouses may enable a fuller picture of what types of responses exist, which interventions may be most beneficial, and what other factors may relate to positive coping, increased resilience and quality of life, such as flexibility, and the nature of the couples' dyadic coping.

All new incoming married patients to the Institute of Radiotherapy at the Tel Aviv (Sourasky) Medical Center from September to January, 2007 will be presented with the request to participate in this research. Overall, we plan to recruit 40 breast and prostate cancer patients and their spouses.

Measures:

1. Demographic and medical questionnaire (adapted to the type of illness).
2. Exposure to trauma. Participants' exposure to possible traumatic events was assessed by The Trauma History Scale created by Pat-Horenczyk in 2004 based on the Posttraumatic Diagnostic Scale (PDS) by Foa, Cashman, Jaycox, and Perry (1997).
3. Posttraumatic Stress Diagnostic Scale (PDS). A self-report assessment that meets all the criteria of the DSM-IV for diagnosis of PTSD developed by Foa, Cashman, Jaycox & Perry, 1997).
4. Depression questionnaire (CESD, The Centre For Epidemiological Studies Depression Scale (CES-D).
5. Flexibility Questionnaire: The Flexibility Scale was developed by Bonanno and Pat-Horenczyk in (2006) and translated into Hebrew.
6. Dyadic coping : The quality of adjustment in the marital relationship will be measured using the Dyadic Adjustment Scale (DAS). This 32 item measure is widely used in clinical and research settings and consists of four subscales: Dyadic Consensus, Dyadic Satisfaction, Dyadic Cohesion and Affectional Expression.
7. Self efficacy: The GSE (General perceived self efficacy scale) was developed by Zeidner, Jerusalem & Schwarzer (1993) and includes 10 items which measure positive self statements with regards to a variety of coping requirements.
8. Ego Resilience: The short 14 item version of Ego-Resiliency Scale was presented in 1996 by Block & Kremen (1996).

Procedure:

Physicians working at the Institute of Radiotherapy at the Tel Aviv (Sourasky) Medical Center will inform all potential participants about the purpose of the study. Those who show interest and match the inclusion criteria will be asked to sign the informed consent with the doctor, who will provide more detailed information. The research assistant will set up a meeting at the Medical Center with the each interested couple (individually with each couple) to fill out the questionnaires. The approximate time for filling out the entire battery is 30 minutes. In order to participate, both patients and their spouses must agree to fill out the questionnaires at the three time points.

In the informed consent it will be specified that participants who may experience distress following the questionnaire or as a result of the research will be offered short individual or couple counseling as needed by the psychosocial staff of the Institute of Radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Dyadic pairs (not necessarily married, but in couples)
* One member of the couple has breast cancer or prostate cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-10; Study Completion 2008-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin W Corn, M.D., Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel